CLINICAL TRIAL: NCT00353886
Title: Retrospective Study of In Utero Antiepileptic Drug Effects in Neurodevelopment
Brief Title: Study of Antiepileptic Drug Effects on Child Development
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Collaborators: GlaxoSmithKline (Industry)
Other Study IDs: RNEAD
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2007-07-23 (Estimated); Status verified 2007-07

CONDITIONS: Epilepsy
Keywords: Retrospective; Epilepsy; Antiepileptic Drugs; Behavioral Development; Intellectual Development
MeSH Terms: conditions — Epilepsy | interventions — Traumeel S

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: TONI-3
Procedure: WRAT-3
Procedure: Connor's Rating Scales PRS & TRS
Procedure: Peabody Picture Vocabulary Test
Procedure: Children's Memory Scale
Procedure: WISC-3
Procedure: Behavioral Assessment System for Children PRS & TRS

SUMMARY:
The specific aim of this study is to determine if in utero exposure produces differential antiepileptic drug (AED) effects on subsequent cognitive abilities and behavioral abnormalities in children

DETAILED DESCRIPTION:
Subject groups will include 120 children (6 - 16 year/old) of women with epilepsy, who were exposed to one of the following anti-epileptic drugs during the mother's pregnancy with that child: Carbamazepine/Tegretol, Valproate/Depakote, and Phenytoin/Dilantin.

In addition to the children, their mother, father and a primary relative of the mother will also be asked participate in the study. Children cannot be enrolled if they were exposed to another known teratogen during their mother's pregnancy other than the target AEDs in monotherapy; if the child has or has had a serious brain injury (e.g. severe head trauma) or serious medical illness (e.g. cancer), which is unrelated to AED exposure and may affect the child's cognitive abilities. Other exclusion criteria include, maternal IQ <70; mother has a progressive brain lesion (e.g. tumor) or mother had serious medical illness or complication during this child's pregnancy, which was unrelated to AED or epilepsy, history or maternal alcohol or drug abuse in past 12 months, and history of child abuse. If possible, the child should be off sympathomimetic medications (e.g. Ritalin) for 24 hours prior to testing if he/she is being treated for ADD or ADHD.

Procedures: The primary test is the IQ (TONI-3) in the children. Additional tests in the children include the Peabody Picture Vocabulary Test -3; WRAT spelling, math & reading subtests; Children's Memory Scale: story memory subtest (immediate, delayed, & delayed recognition subscales); WISC-III coding subtest; Behavioral Assessment System for Children (parent and teacher scales) and the Conner's Rating Scale - (parent and teacher rating scales).

Collected information about the mother includes social and medical factors of the mother, specifically age, type of epilepsy, AED & estimated months exposed and average dose during pregnancy, estimated seizure frequency during pregnancy (by types including status), any other major medical illnesses during pregnancy, primary language, education level and socioeconomic status. The mother will also have an IQ (TONI-3) test.

Collected information about the child include: age, gender, gestational age at birth (i.e. full or pre-term), birth order & # sibs, primary language at home, Birth defects, Hx ADD or ADHD; other major medical illnesses (include perinatal complications); special education requirements of the child; and remedial math or reading requirements of child.

Collected information about the father and primary relative include: age, relationship to mother (for primary relative), primary language, education level, socioeconomic status, any major medical illnesses (especially those which could affect IQ). The relative and father will also have an IQ (TONI-3) test.

ELIGIBILITY:
Inclusion Criteria:

1. Children presently 6-16 years/old who were exposed in utero to monotherapy with carbamazepine, phenytoin, or valproate because their mother had epilepsy and was taking one of these monotherapies while pregnant with the child.
2. In utero exposure should be at least 6 months.
3. Children of the same mother may be enrolled if each child was exposed to a different AED monotherapy (e.g. carbamazepine, phenytoin, or valproate) during their mother's pregnancy.
4. Mother's primary language should be English or Spanish.
5. The mother was 18-35 years of age when the child was born (inclusive).

Exclusion Criteria:

1. Child was exposed to another known teratogen during their mother's pregnancy other than the target AEDs in monotherapy.
2. Child is presently on a centrally active medication other than sympathomimetics (e.g. Ritalin) for ADD or ADHD. Child should be off the sympathomimetic for at least 24 hours prior to testing.
3. Child has or has had a serious brain injury (e.g., severe head trauma) or serious medical illness (e.g., cancer) unrelated to AED exposure, which may affect the child's cognitive abilities.
4. Mother has IQ < 70.
5. Mother has a progressive brain lesion (e.g., tumor).
6. Mother had serious medical illness or complication during this child's pregnancy, which was unrelated to AED or epilepsy.
7. Mother has known history of drug or alcohol abuse within the previous 12 months or has sequelae of drug abuse.
8. There is a known history of child abuse.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2002-09; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Lee, Ph.D., Principal Investigator — Augusta University; Kimford J. Meador, MD, Study Chair — University of Florida
Locations (10):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Boston University, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Case Western Reserve University, Cleveland, Ohio
- University of Aberdeen, Aberdeen, United Kingdom

REFERENCES:
- See also: Related Info — https://web.emmes.com/study/nead/